CLINICAL TRIAL: NCT06024499
Title: A Randomized, Double-blind, Placebo-controlled, Multicenter, Phase 2 Study to Evaluate the Efficacy and Safety of HY209 Gel in Patients With Mild to Moderate Atopic Dermatitis(AD)
Brief Title: Phase 2 Trial of HY209gel in Atopic Dermatitis Patients
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Shaperon (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HY209-AD-02
Record Dates: First submitted 2023-07-24; First posted 2023-09-06 (Actual); Last update posted 2024-04-26 (Actual); Status verified 2023-07

CONDITIONS: Atopic Dermatitis; Atopic Dermatitis Eczema; Atopic Dermatitis of Scalp
MeSH Terms: conditions — Dermatitis, Atopic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: A Randomized, Double-blind, Placebo-controlled Study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- PART 2 High-Dose (Active Comparator): Active group selected for PART1 as a high-dose
  Interventions: Drug: HY209GEL Active
- PART 2 Low-Dose (Active Comparator): Active group selected for PART1 as a Low-dose
  Interventions: Drug: HY209GEL Active
- PART 2 Placebo (Placebo Comparator): Placebo group
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: HY209GEL Active — Selected two among four doses (HY209GEL 0.5% or 1% or 2% or 4%) in PART1
  Arms: PART 2 High-Dose; PART 2 Low-Dose
Other: Placebo — Placebo
  Arms: PART 2 Placebo

SUMMARY:
This is a randomized, double-blind, placebo-controlled, multi-center, phase 2 study in patients with mild to moderate Atopic Dermatitis(AD), which consists of 2 parts.

DETAILED DESCRIPTION:
Part 1 (2 cohorts): Total 33 subjects

* Cohort A: 15 subjects (6 HY209gel 0.5%, 6 HY209gel 1%, and 3 placebo)
* Cohort B: 9 subjects (6 HY209gel 2%, and 3 placebo)
* Cohort C: 9 subjects (6 HY209gel 4%, and 3 placebo)

Part 2 (3 treatment groups): Total 177 subjects

* Low dose of HY209gel: 59 subjects
* High dose of HY209gel: 59 subjects
* Placebo (Vehicle): 59 subjects

Part 1 is a dose-escalation part of HY209gel using lower doses of HY209gel (0.5% and 1%) with escalation (HY209gel 2% and 4%) to evaluate the pharmacokinetics(PK), safety, and tolerability of HY209gel treatment. Escalation to the next dose level will be decided by the Safety Monitoring Committee(SMC) that will review all available safety data of the planned dose level within the timeline specified on SMC charter after all enrolled subjects of each cohort complete 2-week treatment and determine the escalation to the next dose to be safe.

Based on the interim analysis for 4-week safety and efficacy data collected from Part 1, two doses will be selected for use in Part 2, which will enroll up to 177 subjects in 3 treatment arms (59 subjects per treatment arm) to evaluate the efficacy and safety of HY209gel, compared to placebo (vehicle) for 8-week treatment period.

ELIGIBILITY:
Key Inclusion Criteria:

* Male or female subjects aged 18 or older
* Subjects who have a history of AD at least 6 months ago from screening and have been clinically stable for ≥ 1 month
* Subjects with a clinical diagnosis of AD according to the Hanifin and Rajka Criteria by a board certified/eligible dermatologist
* Subjects who have a minimum of 5% and a maximum of 30% of total body surface area (BSA) affected by AD at screening and baseline visits
* Subjects with vIGA score 2 or 3 corresponding to mild to moderate AD at screening and baseline visit
* Subjects should be a literate person who can read the participant information sheet and consent form/questionnaire and understand the language of the participation

Key Exclusion Criteria:

* Subjects who have unstable AD (i.e., remaining clinical stable less than 6 months) or any consistent requirement for any potency topical corticosteroids
* Subjects who have topical treatment with corticosteroids within 2 weeks prior to baseline visit or other topical treatments of the AD area at screening (moisturizers/emollients are allowed)
* Subjects who had systemic treatment with corticosteroids or cyclosporine or other immunosuppressive treatments within 4 weeks prior to baseline visit
* Subjects who had dupilumab or any other biologics within 6 months prior to baseline visit
* Subjects who take any systemic anti-infective or antibiotic treatments within 1 week prior to baseline visit
* Subjects who had ultraviolet irradiation (including photopheresis) within 4 weeks prior to screening
* Subjects who have active malignancy or history of cancer in 5 years prior to screening, except for treated cautions basal cell carcinoma and in situ cervical cancer
* Subjects who have any other skin diseases that would affect the ability to assess the AD
* Subjects who are taking strong CYP3A4 inhibitor or any other concomitant drug that, in the opinion of the PI, may cause interference with the treatment
* Subjects who participated in another drug or device trial within 4 weeks prior to screening...etc

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 210 (Estimated)
Dates: Start 2024-03-01 (Actual); Primary Completion 2025-10-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Percentage change in Eczema Area and Severity Index (EASI) score | at Week 8
  To achieve lower score means disease improvement .

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - Cahaba Dermatology Skin Health Center, Birmingham, Alabama
  - RAOOF MD Dermatology, Encino, California
  - Continental Clinical Solutions, LLC, Towson, Maryland
  - Sadick Dermatology, New York, New York